CLINICAL TRIAL: NCT01247558
Title: Administrative Claims Analysis of Metanx® in Diabetic Peripheral Neuropathy
Status: Completed | Type: Observational
Sponsor: Pamlab, L.L.C. (Industry)
Collaborators: HealthCore, Inc. (Industry)
Responsible Party: Sponsor
Organization: Pamlab, Inc. (Industry)
Other Study IDs: M-006
Record Dates: First submitted 2010-11-17; First posted 2010-11-24 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Diabetic Peripheral Neuropathy (DPN)
Keywords: Metanx®; diabetes; neuropathy; peripheral neurological disorder; peripheral circulation disorder; folic acid; folate; L-methylfolate; vitamin B6; Pyridoxal 5'-phosphate; vitamin B12; methylcobalamin
MeSH Terms: conditions — Diabetes Mellitus | interventions — metanx

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Test Cohort: 100 randomized subjects administered Metanx®
  Interventions: Other: Metanx® (a medical food)
- Control Cohort: 400 subjects with diabetes mellitus meeting the same inclusion and exclusion criteria as the test cohort who have not been treated with Metanx®.
  Interventions: Other: Not treated with Metanx®

INTERVENTIONS:
Other: Metanx® (a medical food) — Patient cohort compliant on Metanx® BID therapy for >120 days
  Groups: Test Cohort
Other: Not treated with Metanx® — Non-treated comparative cohort
  Groups: Control Cohort

SUMMARY:
This study will be an observational cohort study utilizing administrative claims data with 100 patients randomly selected taking Metanx® meeting the inclusion and exclusion criteria and 400 propensity score matched patients meeting the same criteria to serve as a control cohort for analyses. This data includes medical, and pharmacy claims from the HealthCore Integrated Research Database for claims submitted during the time period of 01/01/2002 through 06/30/2007.

DETAILED DESCRIPTION:
The control patients will be matched at a ratio of 4:1 with the Metanx® patients. Covariates used to select the propensity matched patients will include: age; gender; health plan type and region; DCI score; presence/absence of nephropathy; ischemic heart disease; cerebrovascular disease; neoplasm; insulin use; and all-cause health plan costs in the 6-mont pre-index period.

Claims information about patients selected for the study will be followed longitudinally to the end of data availability. This data stream will be used to determine treatment patterns for Metanx®, healthcare resource utilization, and cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pharmacy claims for >120 continuous days of Metanx®. This will be defined as at least a 90-day supply dispensed within the first 120 days post-index. The first pharmacy claim for Metanx® will be the index date.
* Patients must have a diagnosis of diabetes prior to or including the index date.
* Patients must have a diagnosis of a peripheral neurological or a peripheral circulation disorder.
* Patients must have a diagnosis of lower limb ulcer.

Exclusion Criteria:

* Patients will be excluded if they have <18 months of eligibility defined as a minimum of 6 months pre and 12 months post-index eligibility.
* Patients will be excluded if they have taken other L-methylfolate containing products (Deplin®, Cerefolin®, Cerefolin NAC®,Neevo®) or other prescription folic acid combination products with >1mg folic acid.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Diabetes and Peripheral Neuropathy or Peripheral Circulatory Disorder with Lower Limb Ulceration Who Have Been Treated with Metanx® or Not Treated with Metanx®.
  Patients selected for the study will be identified from a review of available medical and pharmacy data during the period from 01/01/2003 to 06/30/2006. The date of the first pharmacy claim of interest within the intake period will be defined as the index date.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
All-Cause Health Plan Costs | 12 months post-index period
  Total healthcare utilization and costs for patients treated with Metanx® will be compared to total healthcare utilization and costs for control patients who did not receive Metanx®. Cost data will be presented as Mean (SD) and median.

SECONDARY OUTCOMES:
Disease-Attributable Resoure Use and Cost | 12 month post-index period
  Disease attributable resource use and costs will be defined as medical claims associated with ICD-9 codes for disease(s) of interest. Total attributable resource use (units) and cost (allowed or paid), if available, will include: pharmacy (medication related to disease of interest); laboratory tests (all claims); office-based encounters and costs; emergency room visits and cost; other outpatient facility (e.g. clinic, home health); in-patient hospitalization; and durable medical equipment.
Demographics of Patients Taking Metanx® | >120 continuous days Metanx® therapy
  Statistical data including age (at index date); gender; comorbidities; prior and concomitant medications; and Metanx® utilization (e.g. dispensing quantity, number of fills, compliance, and persistency) will be collected to provide a descriptive analysis of the typical Metanx® patient characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Wade, RPh, MS, Study Director — HealthCore, Inc.
Locations (1):
- HealthCore, Inc., Wilmington, Delaware, United States